CLINICAL TRIAL: NCT03730766
Title: Analysis of the Impact of Helicobacter Pylori Infection and Eradication on Salivary Microbiome in Adults by 16S Pyrosequencing
Brief Title: Analysis of the Impact of Helicobacter Pylori on Salivary Microbiome in Adults
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hong Lu, MD, Medical Doctor of Division of Gastroenterology and Hepatology of Renji Hospital,Professor of Medicine, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: rjyy20180801
Record Dates: First submitted 2018-11-02; First posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Helicobacter Pylori Infection
Keywords: helicobacter pylori, saliva microbiota
MeSH Terms: interventions — Esomeprazole; Amoxicillin; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bismuth Plus triple Therapy (Experimental): Esomeprazole 20mg bid, Bismuth Potassium Citrate 600mg bid, Amoxicillin 1.0g tid and Metronidazole 0.4g tid for 14 days
  Interventions: Drug: Esomeprazole; Drug: Amoxicillin; Drug: Bismuth Potassium Citrate

INTERVENTIONS:
Drug: Esomeprazole — Proton pump inhibitor
Drug: Amoxicillin — Antibiotics for H. pylori eradication
  Other Names: Metronidazole
Drug: Bismuth Potassium Citrate — Gastric mucosal protective drug with anti-H. pylori effect

SUMMARY:
Helicobacter pylori (H. pylori), a bacteria transmitted from human to human through upper digestive tract as well as fecal-oral transmission, had infected more than half of people around the world. However, the quantity of H. pylori in oral cavity and its influence on oral microbiota remains to be unclear. The aim of the present study was to examine the effects of H. pylori infection as well as its eradication on oral microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Participants with non-ulcer functional dyspepsia or peptic ulcer disease
* Ability and willingness to participate in the study and to sign and give informed consent
* Received both endoscopy and 13C urea breath test (13C-UBT) before enrolled

Exclusion Criteria:

* Less than 18 years old
* With previous gastric surgery
* Major systemic diseases
* Pregnancy or lactation
* Allergy to any of the study drugs Administration of antibiotics, bismuth, antisecretory drugs in 8 weeks prior to inclusion
* The use of antibiotics or PPI within 2 months before the study
* The presence of dental carious or any untreated cavitated carious lesions and oral abscesses

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-11-15 (Estimated); Study Completion 2018-11-20 (Estimated)

PRIMARY OUTCOMES:
Change of saliva microbiota after eradication | Two months after completion of therapy.
  Two months after completion of therapy, saliva microbiota was assessed by 16S rDNA Pyrosequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Lu, M.D., Ph.D., Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ji Y, Liang X, Lu H. Analysis of by high-throughput sequencing: Helicobacter pylori infection and salivary microbiome. BMC Oral Health. 2020 Mar 20;20(1):84. doi: 10.1186/s12903-020-01070-1. PMID 32197614